CLINICAL TRIAL: NCT01685450
Title: Validation of a New Non Invasive Method of Indirect Measurement of the Intracranial Pressure Variations
Brief Title: NIMIP: Non Invasive Measurement of the Intracranial Pressure
Acronym: MINIPIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Echodia SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CHU 0123; 2010-A00266-33
Record Dates: First submitted 2012-08-31; First posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Hydrocephalus
Keywords: Cochlear microphonic potential; non invasive method; indirect measurement; intracranial pressure; adults

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Intracranial pressure (Other)
  Interventions: Device: Echodia® hand-held equipment

INTERVENTIONS:
Device: Echodia® hand-held equipment

SUMMARY:
The intracranial pressure (ICP), defined by the hydrostatic pressure of the cerebrospinal fluid (CSF), is a key parameter for diagnosing and treating several neurosurgical diseases. Continuous ICP monitoring has an important place in neuro-intensive care for patients with severe head trauma and severe meningeal hemorrhage.

Until now the assessment of ICP requires invasive methods, with a pressure transducer either within the ventricular CSF or within the brain parenchyma. The pressure sensor placement is performed in a neurosurgery department. These invasive methods have also disadvantages: highest risk of infections, catheter misplaced, and risk of bleeding. All these justify the development of a non invasive method. The Biophysics Laboratory (School of Medicine of Clermont-Ferrand) described that the intra-labyrinthic pressure (ILP) modify the functional activities of the outer hair cells in the cochlea.

Cochlear activities' recording is non-invasive and technically simple. A probe is gently inserted into the outer portion of the external ear canal.

Anatomical studies showed communication between the subarachnoid spaces and the perilymphatic compartment by the cochlear aqueduct. Thereby, increases in ICP are transferred to increases in intra-cochlear pressure, which is detected as modifications in cochlear activities.

CSF dynamic tests, as constant flow infusion test, are conducted in patients in the diagnosis of the idiopathic adult hydrocephalus syndrome. Artificial CSF is infused through a lumbar needle, into the CSF space at a constant rate, and the corresponding rise in ICP is registered and analyzed.

The objective of this study is to assess prospectively the accuracy and the precision of a new method for non invasive ICP measurement (using cochlear activities) compared with invasive gold standard CSF pressure measurement during CSF dynamic tests.

DETAILED DESCRIPTION:
The purpose of this study is to examine the evolution of the electrophysiological cochlear activity (cochlear microphonic potential, CMP), with a non invasive method, during invasive ICP monitoring. The data analysis will determine relationship between ICP variations and CMP variations.

Patients, from the neurosurgery department, investigated for 'normal pressure' chronic hydrocephalus are involved in CSF dynamic test. This complex protocol, including infusion test and invasive CSF monitoring, is needed in order to confirm the diagnosis. CSF dynamic tests, a socalled 'perfusion test', are performed in an operating theater, the patient had to be awake but sedated. During perfusion test, electrophysiological cochlear activities are measured with a gold tiptrode (Etymotic Research, Elk Grove Village, Ill) gently inserted into the ear canal.

Electrophysiological cochlear activities, so called electrocochleography (ECochG), are a non invasive and totally passive method used in routine in ENT department. The response measured in ECochG is the cochlear microphonic potential (CMP), generated by the outer hair cells following by presenting tone burst at 1kHz. CMP is recorded with the help of an Echodia® hand-held equipment.

Previously animal studies have shown that the phase of CM is sensitive to ICP changes and CM phase shifts exhibit the same time course as those of otoacoustic emissions (DPOAEs).

The phase changes of CM can indeed be used as a non-invasive tool for monitoring intralabyrinthine and intracranial pressures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected chronic hydrocephalus, undergoing a CSF dynamic test (perfusion test)
* Age greater than 18
* Subject provides written informed consent, or consent form signed by a close relative (husband, wife, children, legal guardian),
* Patient covered under French social security or being a beneficiary of such a regime under the terms of the Act of August 9, 2004

Exclusion Criteria:

* refusal to sign a consent form

  * under otoscopy, presence of obstruction of the ear canal with wax (cerumen).
  * Impossibility of electrophysiological measurements (pathophysiological reason)
  * Technical troubles with the device
  * Patient uncovered under French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Cochlear Microphonic Potential | acquisition every minutes during "Cerebrospinal Fluid Dynamic Test time(30-45min)

SECONDARY OUTCOMES:
IntraCranialPressure Variations | every minutes during CerebroSpinal Fluid dynamic test time (30-45min)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SAKKA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France